CLINICAL TRIAL: NCT00927186
Title: Skeletal Histomorphometry in Patients on Teriparatide or Zoledronic Acid Therapy
Brief Title: Effects of Teriparatide or Zoledronic Acid Treatment on Bone in Postmenopausal Osteoporotic Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13032; B3D-US-GHDL (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Results first posted 2012-03-02 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-02

CONDITIONS: Osteoporosis, Post-menopausal
Keywords: osteoporosis; teriparatide; zoledronic acid; histomorphometry; bone biopsy; postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Teriparatide; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriparatide (Experimental)
  Interventions: Drug: Teriparatide
- Zoledronic Acid (Active Comparator)
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Teriparatide — 20 microgram (mcg) subcutaneous (SC) injection per day for 12 months. Placebo intravenous (IV) infusions were given to maintain blind.
  After completing 12 months of treatment, all participants are eligible to participate in an additional 12-month extension.
  Other Names: LY333334; Forteo; Forsteo
  Arms: Teriparatide
Drug: Zoledronic Acid — 5 milligram (mg) intravenous (IV) infusion administered once during 1 year study. Placebo subcutaneous (SC) injections were given to maintain blind.
  After completing 12 months of treatment, all participants are eligible to participate in an additional 12-month extension.
  Arms: Zoledronic Acid

SUMMARY:
The purpose of this study is to investigate how teriparatide or zoledronic acid affects the bone of postmenopausal osteoporotic women after 6 months of treatment as determined by a bone biopsy sample taken from the iliac crest (upper part of the pelvis). After completing 12 months of treatment all participants are eligible to participate in an additional 12-month open label extension.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, postmenopausal women with osteoporosis (no vaginal bleeding for at least 2 years prior to trial entry)
* Free of severe or chronically disabling conditions other than osteoporosis that will impair ability to complete the trial
* Bone mineral density (BMD) T-score of at least -2.5 at the femoral neck, total hip, or lumbar spine (L1-L4, with at least 2 evaluable vertebrae), with or without atraumatic fracture or,
* Bone mineral density (BMD) T-score of at least -1.5 at the femoral neck, or total hip, or lumbar spine (L1-L4, with at least 2 evaluable vertebrae), and either 1 or more atraumatic vertebral fracture(s) or an atraumatic nonvertebral fracture in the opinion of the investigator. Nonvertebral fracture sites allowed are wrist, hip, pelvis, ribs, humerus, clavicle, leg (femur, tibia, and fibula, excluding the ankle).
* Serum calcium, parathyroid hormone (PTH), alkaline phosphatase must be within normal reference range

Exclusion Criteria:

* Have an increased risk of osteosarcoma (bone tumor); this includes Paget's disease of bone, a previous bone tumor, or radiation involving the skeleton
* Are allergic or cannot tolerate teriparatide or zoledronic acid or any of their ingredients or components
* Are allergic to tetracycline
* Have a history of exposure to tetracycline therapy in the 3 months prior to trial entry
* Have participated in a prior PTH clinical trial or received prior treatment with teriparatide, PTH, or other related medications
* Have a vitamin D level below 10 nanogram/milliliter (ng/mL)
* Have a condition that could possibly put one at risk for an adverse event due to the bone biopsy procedure (e.g. bleeding disorder)
* Have undergone two previous iliac crest bone biopsies (one in each iliac crest)
* Have taken any intravenous (IV) osteoporosis medication
* Have taken other oral osteoporosis medications and have not been off of them for a specific period of time before trial entry
* Have a history of certain cancers in the 5 years prior to trial entry
* Have active liver disease
* Have significantly impaired kidney function
* Currently have active or suspected diseases that affect the bones, other than osteoporosis
* Have active or recent history of significant gastrointestinal (stomach or intestinal) disorders
* Have been treated with certain glucocorticoids for more than 30 days in the past 1 year prior to trial entry

Ages: 55 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Haverstraw, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sainte-Foy, Quebec

REFERENCES:
- [Derived] Dempster DW, Zhou H, Recker RR, Brown JP, Bolognese MA, Recknor CP, Kendler DL, Lewiecki EM, Hanley DA, Rao SD, Miller PD, Woodson GC 3rd, Lindsay R, Binkley N, Alam J, Ruff VA, Gallagher ER, Taylor KA. A Longitudinal Study of Skeletal Histomorphometry at 6 and 24 Months Across Four Bone Envelopes in Postmenopausal Women With Osteoporosis Receiving Teriparatide or Zoledronic Acid in the SHOTZ Trial. J Bone Miner Res. 2016 Jul;31(7):1429-39. doi: 10.1002/jbmr.2804. Epub 2016 Mar 8. PMID 26841258

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a Phase 4, multicenter, randomized, stratified, double-blind, active comparator-controlled study with the primary endpoint at 6 months. Following the bone biopsy visit at 6 months, the study became open label for an additional 6 months. All participants who complete 12 months of treatment are eligible for an additional 12-month extension.
Period: 12 Months Primary Study
Arm/Group | Teriparatide | Zoledronic Acid
Started | 34 | 35
Completed 6 Months Double Blind Phase | 28 | 31
Completed | 27 | 31
Not Completed | 7 | 4
Not completed — Adverse Event | 5 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: 12 - 24 Months Extension Treatment
Arm/Group | Teriparatide | Zoledronic Acid
Started | 10 (Not all participants who completed 12 months of primary study chose to enter 12-month extension.) | 11 (Not all participants who completed 12 months of primary study chose to enter 12-month extension.)
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Zoledronic Acid | Total
Number analyzed (Participants) | 34 | 35 | 69
Age Continuous [Mean (Standard Deviation); unit: years] | 65.49 (6.93) | 64.20 (5.96) | 64.84 (6.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 35 | 69
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 1 | 2
  White | 33 | 34 | 67
Region of Enrollment [Number; unit: participants]
  United States | 21 | 25 | 46
  Canada | 13 | 10 | 23
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 159.28 (5.92) | 160.00 (7.38) | 159.64 (6.66)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 61.25 (9.21) | 64.75 (11.66) | 63.03 (10.60)
Pulse [Mean (Standard Deviation); unit: beats per minute (bpm)] | 67.41 (7.15) | 70.60 (8.79) | 69.03 (8.13)
Blood Pressure - Systolic [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] | 125.71 (16.19) | 122.49 (16.25) | 124.07 (16.18)
Blood Pressure - Diastolic [Mean (Standard Deviation); unit: mmHg] | 74.79 (8.24) | 73.97 (10.15) | 74.38 (9.20)
Alcohol Use [Number; unit: participants]
  Yes | 21 | 17 | 38
  No | 13 | 18 | 31
Tobacco Use [Number; unit: participants]
  Yes | 5 | 5 | 10
  No | 29 | 30 | 59
Caffeine or Xanthine Use [Number; unit: participants]
  Yes | 29 | 30 | 59
  No | 5 | 5 | 10
Previous Osteoporosis Therapy [Number; unit: participants]
  Yes | 17 | 21 | 38
  No | 17 | 14 | 31
Fracture Status [Number; unit: participants] — Yes means a participant has already had fracture before study entry.
  participants
    Yes | 14 | 17 | 31
    No | 20 | 18 | 38
Lumbar Spine T-Score [Mean (Standard Deviation); unit: T-Score] — The T-score at lumbar spine is a comparison of a participant's bone mineral density (BMD) to that of the mean BMD for a healthy population of women at peak bone mass (30 years). A normal T-score has a value of -1.0 or higher. Osteoporosis is defined as a T-score of -2.5 or lower, meaning a bone mineral density that is two and a half standard deviations below the mean BMD of a healthy population of women at peak bone mass (30 years).
  T-Score | -2.79 (0.83) | -2.93 (0.75) | -2.86 (0.79)
Femoral Neck T-Score [Mean (Standard Deviation); unit: T-Score] — The T-score at femoral neck is a comparison of a participant's bone mineral density (BMD) to that of the mean BMD for a healthy population of women at peak bone mass (30 years). A normal T-score has a value of -1.0 or higher. Osteoporosis is defined as a T-score of -2.5 or lower, meaning a bone mineral density that is two and a half standard deviations below the mean BMD of a healthy population of women at peak bone mass (30 years).
  T-Score | -2.25 (0.68) | -2.29 (0.74) | -2.27 (0.70)
Total Hip T-Score [Mean (Standard Deviation); unit: T-Score] — The T-score at total hip is a comparison of a participant's bone mineral density (BMD) to that of the mean BMD for a healthy population of women at peak bone mass (30 years). A normal T-score has a value of -1.0 or higher. Osteoporosis is defined as a T-score of -2.5 or lower, meaning a bone mineral density that is two and a half standard deviations below the mean BMD of a healthy population of women at peak bone mass (30 years).
  T-Score | -1.78 (0.78) | -1.88 (0.91) | -1.83 (0.84)
Serum Procollagen Type I N-Terminal Propeptide (PINP) [Mean (Standard Deviation); unit: microgram/Liter (µg/L)] — A measure of bone formation.
  microgram/Liter (µg/L) | 49.18 (18.28) | 52.88 (19.43) | 51.03 (18.81)
Serum Carboxyterminal Cross-Linking Telopeptide of Collagen Type I (CTX) [Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)] — A measure of bone resorption.
  nanogram/milliliter (ng/mL) | 0.43 (0.23) | 0.42 (0.19) | 0.43 (0.21)
Serum Osteocalcin [Mean (Standard Deviation); unit: microgram/Liter (µg/L)] — A measure of osteoblast function.
  microgram/Liter (µg/L) | 25.05 (8.37) | 24.92 (8.53) | 24.98 (8.39)

OUTCOME MEASURES:

1. Primary Outcome: Mineralizing Surface/Bone Surface (MS/BS) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 6 Months
Description: MS/BS in CC is a measure of the proportion of BS on which new mineralized bone is deposited at the time of tetracycline (T) labeling and is calculated as sum of total extent of double label (DL) plus half the extent of single label (SL) divided by BS. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in the biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under a microscope. DL indicates active bone formation, SL or no label (NL) suggests suppression of bone formation.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: percentage of surface
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
percentage of surface | 5.60 (10.20) [3.00 to 11.75] | 0.16 (2.62) [0.00 to 0.58]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — The pre-specified significance level 0.05 was used

2. Secondary Outcome: Mineralizing Surface/Bone Surface (MS/BS) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 24 Months
Description: as for outcome 1
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had MS/BS analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: percentage of surface
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 9
percentage of surface | 3.00 [1.49 to 4.58] | 0.07 [0.00 to 0.42]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Mineralizing Surface/Bone Surface(MS/BS) in the Endocortical Compartment (EC) of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: MS/BS in EC is a measure of the proportion of BS on which new mineralized bone is deposited at the time of tetracycline (T) labeling and is calculated as sum of total extent of double label (DL) plus half the extent of single label (SL) divided by BS. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in the biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under a microscope. DL indicates active bone formation, SL or no label (NL) suggests suppression of bone formation.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had MS/BS analysis of the EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: percentage of surface
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 29
percentage of surface
  6 months (n=23, 29) | 18.64 [9.25 to 21.96] | 0.30 [0.00 to 0.84]
  24 months (n=9, 8) | 5.82 [3.10 to 7.08] | 0.00 [0.00 to 0.91]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — P-value is for 24 months

4. Secondary Outcome: Activation Frequency (Ac.f) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 6 Months
Description: Ac.f in CC represents the frequency of activation of new remodeling cycles on BS (bone formation rate [BFR]/BS divided by wall thickness) and is expressed in units of new cycles per unit of time. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 micrometer (µm)/day or counted as missing.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: new cycles/year
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
new cycles/year
  DL and NL (n=28, 28) | 0.37 [0.17 to 0.82] | 0.01 [0.00 to 0.04]
  DL, Imputed SL (ISL) and NL (n=28, 30) | 0.37 [0.17 to 0.82] | 0.01 [0.00 to 0.03]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

5. Secondary Outcome: Activation Frequency (Ac.f) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 24 Months
Description: Ac.f in CC represents the frequency of activation of new remodeling cycles on the bone surface (BFR/BS divided by wall thickness) and is expressed in units of new cycles per unit of time. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had Ac.f analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: new cycles/year
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 9
new cycles/year
  DL and NL (n=9, 6) | 0.19 [0.10 to 0.20] | 0.00 [0.00 to 0.02]
  DL, Imputed SL (ISL) and NL (n=10, 9) | 0.18 [0.08 to 0.20] | 0.00 [0.00 to 0.02]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

6. Secondary Outcome: Activation Frequency (Ac.f) in the Endocortical Compartment (EC) of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: Ac.f in EC represents the frequency of activation of new remodeling cycles on the bone surface (BFR/BS divided by wall thickness) and is expressed in units of new cycles per unit of time. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had Ac.f analysis of the EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: new cycles/year
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 29
new cycles/year
  DL and NL at 6 Months (n=23, 20) | 0.83 [0.49 to 1.09] | 0.00 [0.00 to 0.07]
  DL, Imputed SL (ISL) and NL at 6 Months (n=23, 29) | 0.83 [0.49 to 1.09] | 0.01 [0.00 to 0.04]
  DL and NL at 24 Months (n=8, 7) | 0.25 [0.18 to 0.31] | 0.00 [0.00 to 0.07]
  DL, ISL and NL at 24 Months (n=9, 8) | 0.24 [0.14 to 0.29] | 0.00 [0.00 to 0.04]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 6 months
Statistical Analysis 3: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 24 months
Statistical Analysis 4: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 24 months

7. Secondary Outcome: Bone Formation Rate (BFR) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 6 Months
Description: BFR in CC is the volume of mineralized bone formed per unit surface bone per unit time (cubic millimeter/square millimeter/year [mm³/mm²/year]); calculated as mineral apposition rate (MAR) times MS/BS. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: mm³/mm²/year
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
mm³/mm²/year
  DL and NL (n=28, 28) | 0.0116 (0.0666) [0.0051 to 0.0265] | 0.0002 (0.0220) [0.0000 to 0.0010]
  DL, ISL and NL (n=28, 30) | 0.0116 [0.0051 to 0.0265] | 0.0002 [0.0000 to 0.0010]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

8. Secondary Outcome: Bone Formation Rate (BFR) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 24 Months
Description: BFR in CC is the volume of mineralized bone formed per unit surface bone per unit time (mm³/mm²/year); calculated as MAR times MS/BS. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had BFR analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: mm³/mm²/year
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 9
mm³/mm²/year
  DL and NL (n=9, 6) | 0.0057 [0.0033 to 0.0061] | 0.0000 [0.0000 to 0.0005]
  DL, Imputed SL (ISL) and NL (n=10, 9) | 0.0057 [0.0022 to 0.0061] | 0.0001 [0.0000 to 0.0005]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

9. Secondary Outcome: Bone Formation Rate (BFR) in the Endocortical Compartment (EC) of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: BFR in EC is the volume of mineralized bone formed per unit surface bone per unit time (mm³/mm²/year); calculated as MAR times MS/BS. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had BFR analysis of EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: mm³/mm²/year
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 29
mm³/mm²/year
  DL and NL at 6 Months (n=23, 20) | 0.0307 [0.0182 to 0.0411] | 0.0000 [0.0000 to 0.0022]
  DL, Imputed SL (ISL) and NL at 6 Months (n=23, 29) | 0.0307 [0.0182 to 0.0411] | 0.0003 [0.0000 to 0.0014]
  DL and NL at 24 Months (n=8, 7) | 0.0093 [0.0064 to 0.0109] | 0.0000 [0.0000 to 0.0027]
  DL, ISL and NL at 24 Months (n=9, 8) | 0.0090 [0.0049 to 0.0100] | 0.0000 [0.0000 to 0.0016]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 6 months
Statistical Analysis 3: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 24 months
Statistical Analysis 4: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 24 months

10. Secondary Outcome: Mineral Apposition Rate (MAR) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 6 Months
Description: MAR in CC is a measure of the linear rate of production of mineralized bone matrix by osteoblasts and is measured by the mean distance between two consecutive T labels divided by the time interval. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: micrometer (µm)/day
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
micrometer (µm)/day
  DL and NL (n=28, 28) | 0.56 (0.10) [0.48 to 0.62] | 0.35 (0.10) [0.00 to 0.51]
  DL, ISL and NL (n=28, 30) | 0.56 [0.48 to 0.62] | 0.33 [0.00 to 0.51]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

11. Secondary Outcome: Mineral Apposition Rate (MAR) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 24 Months
Description: MAR in CC is a measure of the linear rate of production of mineralized bone matrix by osteoblasts and is measured by the mean distance between two consecutive labels divided by the time interval. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had MAR analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: micrometer (µm)/day
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 9
micrometer (µm)/day
  DL and NL (n=9, 6) | 0.44 [0.40 to 0.52] | 0.00 [0.00 to 0.34]
  DL, Imputed SL (ISL) and NL (n=10, 9) | 0.43 [0.37 to 0.52] | 0.30 [0.00 to 0.30]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.020, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

12. Secondary Outcome: Mineral Apposition Rate (MAR) in the Endocortical Compartment (EC) of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: MAR in EC is a measure of the linear rate of production of mineralized bone matrix by osteoblasts and is measured by the mean distance between two consecutive labels divided by the time interval. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had MAR analysis of the EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: micrometer (µm/day)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 29
micrometer (µm/day)
  DL and NL at 6 Months (n=23, 20) | 0.50 [0.43 to 0.56] | 0.00 [0.00 to 0.41]
  DL, Imputed SL (ISL) and NL at 6 Months (n=23, 29) | 0.50 [0.43 to 0.56] | 0.30 [0.00 to 0.30]
  DL and NL at 24 Months (n=8, 7) | 0.43 [0.38 to 0.50] | 0.00 [0.00 to 0.44]
  DL, ISL and NL at 24 Months (n=9, 8) | 0.42 [0.37 to 0.45] | 0.00 [0.00 to 0.37]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 6 months
Statistical Analysis 3: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.039, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 24 months
Statistical Analysis 4: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.025, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 24 months

13. Secondary Outcome: Adjusted Apposition Rate (Aj.AR) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 6 Months
Description: Aj.AR in CC is MAR averaged over the entire osteoid surface and in a steady state is an estimate of the mean rate of matrix apposition. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: µm/day
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
µm/day
  DL and NL (n=28, 28) | 0.34 (0.22) [0.15 to 0.51] | 0.02 (0.17) [0.00 to 0.06]
  DL, ISL and NL (n=28, 30) | 0.34 [0.15 to 0.51] | 0.02 [0.00 to 0.07]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

14. Secondary Outcome: Adjusted Apposition Rate (Aj.AR) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 24 Months
Description: as for outcome 13
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had Aj.AR analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: micrometer (µm)/day
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 9
micrometer (µm)/day
  DL and NL (n=9, 6) | 0.13 [0.07 to 0.32] | 0.00 [0.00 to 0.13]
  DL, Imputed SL (ISL) and NL (n=10, 9) | 0.12 [0.07 to 0.32] | 0.02 [0.00 to 0.03]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.050, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.016, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

15. Secondary Outcome: Adjusted Apposition Rate (Aj.AR) in the Endocortical Compartment (EC) of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: Aj.AR in EC is MAR averaged over the entire osteoid surface and in a steady state is an estimate of the mean rate of matrix apposition. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had Aj.AR analysis of the EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: micrometer (µm)/day
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 29
micrometer (µm)/day
  DL and NL at 6 Months (n=23, 20) | 0.41 [0.34 to 0.57] | 0.00 [0.00 to 0.05]
  DL, Imputed SL (ISL) and NL at 6 Months (n=23, 29) | 0.41 [0.34 to 0.57] | 0.03 [0.00 to 0.16]
  DL and NL at 24 Months (n=8, 7) | 0.35 [0.25 to 0.45] | 0.00 [0.00 to 0.12]
  DL, ISL and NL at 24 Months (n=9, 8) | 0.32 [0.19 to 0.45] | 0.00 [0.00 to 0.11]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 6 months
Statistical Analysis 3: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 24 months
Statistical Analysis 4: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 24 months

16. Secondary Outcome: Mineralization Lag Time (Mlt) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 6 Months
Description: Mlt in CC is the period between deposition and subsequent mineralization of osteoid. Mlt is calculated as Osteoid Thickness (O.Th) divided by Aj.AR. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
day
  DL and NL (n=28, 16) | 13.63 [11.22 to 29.22] | 75.72 [26.84 to 193.78]
  DL, ISL and NL (n=28, 18) | 13.63 [11.22 to 29.22] | 75.72 [24.99 to 215.85]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

17. Secondary Outcome: Mineralization Lag Time (Mlt) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 24 Months
Description: Mlt in CC is the period between deposition and subsequent mineralization of osteoid. Mlt is calculated as O.Th divided by Aj.AR. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had Mlt analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 5
day
  DL and NL (n=9, 2) | 38.84 [22.81 to 57.02] | 45.67 [37.70 to 53.65]
  DL, Imputed SL (ISL) and NL (n=10, 5) | 45.33 [22.81 to 81.83] | 128.37 [53.65 to 169.31]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.906, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.159, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

18. Secondary Outcome: Mineralization Lag Time (Mlt) in the Endocortical Compartment (EC) of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: Mlt in EC is the period between deposition and subsequent mineralization of osteoid. Mlt is calculated as O.Th divided by Aj.AR. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had Mlt analysis of the EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 15
day
  DL and NL at 6 Months (n=23, 6) | 12.63 [9.03 to 17.46] | 26.97 [24.61 to 72.03]
  DL, Imputed SL (ISL) and NL at 6 Months (n=23, 15) | 12.63 [9.03 to 17.46] | 26.70 [19.84 to 47.31]
  DL and NL at 24 Months (n=8, 2) | 15.67 [10.56 to 22.99] | 42.86 [23.50 to 62.23]
  DL, ISL and NL at 24 Months (n=9, 3) | 17.04 [11.97 to 23.37] | 29.03 [23.50 to 62.23]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.049, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 6 months
Statistical Analysis 3: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.151, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 24 months
Statistical Analysis 4: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.196, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 24 months

19. Secondary Outcome: Osteoid Maturation Time (Omt) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 6 Months
Description: Omt in CC is the period between the onset of deposition and onset of mineralization of a given amount of osteoid. Omt is calculated as O.Th divided by MAR. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
day
  DL and NL (n=28, 16) | 9.99 [8.39 to 10.74] | 9.05 [7.83 to 10.76]
  DL, ISL and NL (n=28, 18) | 9.99 [8.39 to 10.74] | 9.05 [7.97 to 10.80]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.502, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.597, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

20. Secondary Outcome: Osteoid Maturation Time (Omt) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 24 Months
Description: as for outcome 19
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had Omt analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 5
day
  DL and NL (n=9, 2) | 13.42 [11.62 to 13.72] | 17.38 [13.92 to 20.84]
  DL, Imputed SL (ISL) and NL (n=10, 5) | 13.52 [11.62 to 13.81] | 13.92 [13.26 to 18.98]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.077, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.358, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

21. Secondary Outcome: Osteoid Maturation Time (Omt) in the Endocortical Compartment (EC) of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: Omt in EC is the period between the onset of deposition and onset of mineralization of a given amount of osteoid. Omt is calculated as O.Th divided by MAR. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 and 24 Months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had Omt analysis of the EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 15
day
  DL and NL at 6 Months (n=23, 6) | 10.57 [9.67 to 11.06] | 11.27 [9.62 to 12.80]
  DL, Imputed SL (ISL) and NL at 6 Months (n=23, 15) | 10.57 [9.67 to 11.06] | 11.34 [9.92 to 16.34]
  DL and NL at 24 Months (n=8, 2) | 12.30 [9.86 to 16.61] | 14.94 [12.12 to 17.76]
  DL, ISL and NL at 24 Months (n=9, 3) | 13.03 [10.64 to 16.18] | 12.12 [9.54 to 17.76]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.647, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.120, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 6 months
Statistical Analysis 3: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.695, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 24 months
Statistical Analysis 4: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 24 months

22. Secondary Outcome: Total Formation Period (Tt.FP) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 6 Months
Description: Tt.FP in CC is a measure of bone formation and is calculated as wall thickness divided by Aj.AR. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: year
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
year
  DL and NL (n=28, 16) | 0.24 [0.16 to 0.50] | 1.46 [0.44 to 3.10]
  DL, ISL and NL (n=28, 18) | 0.24 [0.16 to 0.50] | 1.46 [0.44 to 3.49]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

23. Secondary Outcome: Total Formation Period (Tt.FP) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 24 Months
Description: as for outcome 22
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had Tt.FP analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: year
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 5
year
  DL and NL (n=9, 2) | 0.60 [0.31 to 1.12] | 0.51 [0.39 to 0.63]
  DL, Imputed SL (ISL) and NL (n=10, 5) | 0.68 [0.31 to 1.15] | 2.62 [0.63 to 2.82]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.198, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

24. Secondary Outcome: Total Formation Period (Tt.FP) in the Endocortical Compartment (EC) of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: Tt.FP in EC is a measure of bone formation and is calculated as wall thickness divided by Aj.AR. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had Tt.FP analysis of the EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: year
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 15
year
  DL and NL at 6 Months (n=23, 6) | 0.24 [0.17 to 0.30] | 0.43 [0.30 to 1.62]
  DL, Imputed SL (ISL) and NL at 6 Months (n=23, 15) | 0.24 [0.17 to 0.30] | 0.54 [0.32 to 1.37]
  DL and NL at 24 Months (n=8, 2) | 0.27 [0.22 to 0.43] | 0.62 [0.38 to 0.86]
  DL, ISL and NL at 24 Months (n=9, 3) | 0.31 [0.22 to 0.50] | 0.86 [0.38 to 0.89]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.022, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 6 months
Statistical Analysis 3: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.151, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 24 months
Statistical Analysis 4: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.139, Wilcoxon (Mann-Whitney) — -value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 24 months

25. Secondary Outcome: Active Formation Period (a.FP) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 6 Months
Description: a. FP in CC is the mean time required to rebuild a new bone structural unit, calculated as wall thickness divided by MAR. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: year
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
year
  DL and NL (n=28, 16) | 0.15 [0.14 to 0.17] | 0.16 [0.15 to 0.19]
  DL, ISL and NL (n=28, 18) | 0.15 [0.14 to 0.17] | 0.16 [0.15 to 0.21]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.154, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.052, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

26. Secondary Outcome: Active Formation Period (a.FP) in the Cancellous Compartment (CC) of Iliac Crest Bone Biopsies at 24 Months
Description: as for outcome 25
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had a.FP analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: year
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 5
year
  DL and NL (n=9, 2) | 0.19 [0.17 to 0.22] | 0.19 [0.14 to 0.25]
  DL, Imputed SL (ISL) and NL (n=10, 5) | 0.19 [0.17 to 0.22] | 0.25 [0.24 to 0.27]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.906, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL)
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.159, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL)

27. Secondary Outcome: Active Formation Period (a.FP) in the Endocortical Compartment (EC) of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: a. FP in EC is the mean time required to rebuild a new bone structural unit, calculated as wall thickness divided by MAR. Participants were given T for two 3 day-periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation. SL cases were imputed to a value of 0.3 µm/day or counted as missing.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had a.FP analysis of the EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: year
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 15
year
  DL and NL at 6 Months (n=23, 6) | 0.20 [0.17 to 0.22] | 0.20 [0.16 to 0.25]
  DL, Imputed SL (ISL) and NL at 6 Months (n=23, 15) | 0.20 [0.17 to 0.22] | 0.28 [0.21 to 0.32]
  DL and NL at 24 Months (n=8, 2) | 0.23 [0.21 to 0.26] | 0.22 [0.20 to 0.25]
  DL, ISL and NL at 24 Months (n=9, 3) | 0.24 [0.21 to 0.27] | 0.25 [0.20 to 0.29]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.979, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 6 months
Statistical Analysis 3: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.695, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL) and no labels (NL) at 24 months
Statistical Analysis 4: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.853, Wilcoxon (Mann-Whitney) — P-value is for double labels (DL), imputed single labels (ISL) and no labels (NL) at 24 months

28. Secondary Outcome: Percent of Single or Double Tetracycline Labels Per Bone Surface (sLS/BS), (dLS/BS) in the Cancellous Compartment of Iliac Crest Bone Biopsies at 6 Months
Description: The percent of single or double tetracycline labels per bone surface (sLS/BS, dLS/BS) in the cancellous compartment. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: percentage of tetracycline labels
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
percentage of tetracycline labels
  sLS/BS | 3.19 (2.85) [1.58 to 4.86] | 0.02 (1.70) [0.00 to 0.38]
  dLS/BS | 4.13 (8.90) [2.14 to 8.88] | 0.07 (1.78) [0.00 to 0.30]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for sLS/BS
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for dLS/BS

29. Secondary Outcome: Percent of Single or Double Tetracycline Labels Per Bone Surface (sLS/BS), (dLS/BS) in the Cancellous Compartment of Iliac Crest Bone Biopsies at 24 Months
Description: as for outcome 28
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had sLS/BS and dLS/BS analysis of the cancellous compartment at 24 months.
Measure: Median (Inter-Quartile Range); unit: percentage of tetracycline labels
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 9
percentage of tetracycline labels
  sLS/BS | 2.25 [1.27 to 2.90] | 0.15 [0.00 to 0.42]
  dLS/BS | 1.69 [0.41 to 3.69] | 0.00 [0.00 to 0.00]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney) — P-value is for sLS/BS
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney) — P-value is for dLS/BS

30. Secondary Outcome: Percent of Single or Double Tetracycline Labels Per Bone Surface (sLS/BS), (dLS/BS) in the Endocortical Compartment of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: The percent of single or double tetracycline labels per bone surface (sLS/BS, dLS/BS) in the endocortical compartment. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had sLS/BS and dLS/BS analysis of the endocortical compartment at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: percentage of tetracycline labels
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 29
percentage of tetracycline labels
  sLS/BS at 6 months (n=23, 29) | 5.56 [3.42 to 8.06] | 0.25 [0.00 to 1.42]
  dLS/BS at 6 months (n=23, 29) | 13.46 [6.04 to 18.68] | 0.00 [0.00 to 0.00]
  sLS/BS at 24 months (n=9, 8) | 3.75 [3.16 to 5.69] | 0.00 [0.00 to 1.12]
  dLS/BS at 24 months (n=9, 8) | 2.77 [0.95 to 2.98] | 0.00 [0.00 to 0.35]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for sLS/BS at 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for dLS/BS at 6 months
Statistical Analysis 3: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney) — P-value is for sLS/BS at 24 months
Statistical Analysis 4: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney) — P-value is for dLS/BS at 24 months

31. Secondary Outcome: Number of Samples With Single or Double Tetracycline Labels, Single and Double Labels, or No Tetracycline Labels in the Cancellous Compartment of Iliac Crest Bone Biopsies at 6 Months
Description: Number of samples with single or double tetracycline labels, both single and double labels, or no labels in the cancellous compartment were compared between teriparatide and zoledronic acid treated participants. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Number; unit: samples
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
samples
  No Label | 0 | 12
  Single Label Only | 0 | 2
  Double Label Only | 0 | 3
  Single and Double Label | 28 | 13
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is a comparison of "No Label" vs. "Single, Double, Single and Double Label"

32. Secondary Outcome: Number of Samples With Single or Double Tetracycline Labels, Single and Double Labels, or No Tetracycline Labels in the Cancellous Compartment of Iliac Crest Bone Biopsies at 24 Months
Description: as for outcome 31
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy of the cancellous compartment at 24 months.
Measure: Number; unit: samples
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 9
samples
  No Label | 0 | 4
  Single Label Only | 1 | 3
  Double Label Only | 0 | 0
  Single and Double Label | 9 | 2
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.033, Fisher Exact — P-value is a comparison of "No Label" vs. "Single, Double, Single and Double Label"

33. Secondary Outcome: Number of Samples With Single or Double Tetracycline Labels, Single and Double Labels, or No Tetracycline Labels in the Endocortical Compartment of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: Number of samples with single or double tetracycline labels, both single and double labels, or no labels in the endocortical compartment were compared between teriparatide and zoledronic acid treated participants. Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy of the endocortical compartment at 6 and 24 months.
Measure: Number; unit: samples
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 29
samples
  No Label at 6 months (n=23, 29) | 0 | 14
  Single Label Only at 6 months (n=23, 29) | 0 | 9
  Double Label Only at 6 months (n=23, 29) | 0 | 0
  Single and Double Label at 6 months (n=23, 29) | 23 | 6
  No Label at 24 months (n=9, 8) | 0 | 5
  Single Label Only at 24 months (n=9, 8) | 1 | 1
  Double Label Only at 24 months (n=9, 8) | 0 | 0
  Single and Double Label at 24 months (n=9, 8) | 8 | 2
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is a comparison of "No Label" vs. "Single, Double, Single and Double Label" at 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.009, Fisher Exact — P-value is a comparison of "No Label" vs. "Single, Double, Single and Double Label" at 24 months

34. Secondary Outcome: Average Length of Tetracycline Double Labels in the Cancellous Compartment of Iliac Crest Bone Biopsies at 6 Months
Description: The length of tetracycline double labels is a measure of the extent of bone formation in the cancellous compartment within individual remodeling units and is measured in millimeters (mm). Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: millimeter (mm)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 16
millimeter (mm) | 0.35 (0.08) [0.28 to 0.38] | 0.24 (0.08) [0.19 to 0.30]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

35. Secondary Outcome: Average Length of Tetracycline Double Labels in the Cancellous Compartment of Iliac Crest Bone Biopsies at 24 Months
Description: as for outcome 34
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had length of tetracycline double labels analysis of the cancellous compartment at 24 months.
Measure: Median (Inter-Quartile Range); unit: millimeter (mm)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 9 | 2
millimeter (mm) | 0.23 [0.22 to 0.29] | 0.29 [0.19 to 0.38]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.906, Wilcoxon (Mann-Whitney)

36. Secondary Outcome: Average Length of Tetracycline Double Labels in the Endocortical Compartment of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: The length of tetracycline double labels is a measure of the extent of bone formation in the endocortical compartment within individual remodeling units and is measured in millimeters (mm). Participants were given T for two 3-day periods, 14 days apart. T fluoresces under certain light and temporarily binds to new bone. New bone in biopsy is seen as the amount of bone between 2 fluorescently T labeled lines under microscope. DL indicates active bone formation, SL or NL suggests suppression of bone formation.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had length of tetracycline double labels analysis of the endocortical compartment at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: millimeter (mm)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 6
millimeter (mm)
  6 months (n=23, 6) | 0.34 [0.27 to 0.39] | 0.30 [0.24 to 0.39]
  24 months (n=8, 2) | 0.27 [0.24 to 0.43] | 0.30 [0.24 to 0.36]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.536, Wilcoxon (Mann-Whitney) — P-value is for 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.896, Wilcoxon (Mann-Whitney) — P-value is for 24 months

37. Secondary Outcome: Percentage of Osteoid Volume (OV)/Bone Volume (BV) in the Cancellous Compartment of Iliac Crest Bone Biopsies at 6 Months
Description: Osteoid volume (OV) in the cancellous compartment is the percent of a given volume of bone tissue that consists of unmineralized bone (osteoid).
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: percentage of volume
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
percentage of volume | 1.32 (1.47) [0.81 to 2.13] | 0.24 (0.76) [0.08 to 0.49]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

38. Secondary Outcome: Percentage of Osteoid Volume (OV)/Bone Volume (BV) in the Cancellous Compartment of Iliac Crest Bone Biopsies at 24 Months
Description: as for outcome 37
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had OV/BV analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: percentage of volume
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 9
percentage of volume | 1.33 [0.89 to 1.56] | 0.18 [0.05 to 0.23]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

39. Secondary Outcome: Percentage of Osteoid Surface (OS)/Bone Surface (BS) in the Cancellous Compartment of Iliac Crest Bone Biopsies at 6 Months
Description: Osteoid surface (OS) in the cancellous compartment is the fraction (%) of the entire trabecular bone surface that is covered by osteoid.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: percentage of surface
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
percentage of surface | 11.34 (8.35) [6.58 to 16.52] | 2.51 (4.84) [1.27 to 4.58]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

40. Secondary Outcome: Percentage of Osteoid Surface (OS)/Bone Surface (BS) in the Cancellous Compartment of Iliac Crest Bone Biopsies at 24 Months
Description: as for outcome 39
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had OS/BS analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: percentage of surface
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 9
percentage of surface | 11.19 [7.23 to 13.14] | 1.26 [0.72 to 2.89]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney)

41. Secondary Outcome: Percentage of Osteoid Surface (OS)/Bone Surface (BS) in the Endocortical Compartment of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: Osteoid surface (OS) in the endocortical compartment is the fraction (%) of the entire trabecular bone surface that is covered by osteoid.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had OS/BS analysis of the EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: percentage of surface
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 29
percentage of surface
  6 months (n=23, 29) | 16.33 [13.57 to 24.34] | 1.87 [1.08 to 3.99]
  24 months (n=9, 8) | 7.48 [6.39 to 10.10] | 1.55 [1.19 to 3.47]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney) — P-value is for 24 months

42. Secondary Outcome: Osteoid Thickness (OTh.) in the Cancellous Compartment of Iliac Crest Bone Biopsies at 6 Months
Description: Osteoid thickness (OTh.) in the cancellous compartment is a measure of the average thickness of osteoid seams.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: micrometer (µm)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
micrometer (µm) | 4.92 (1.38) [4.29 to 6.68] | 3.77 (1.10) [3.51 to 4.22]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

43. Secondary Outcome: Osteoid Thickness (OTh.) in the Cancellous Compartment of Iliac Crest Bone Biopsies at 24 Months
Description: Osteoid thickness (OTh.) in the cancellous compartment is a measure of the average thickness of osteoid seams.
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had OTh. analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: micrometer (µm)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 9
micrometer (µm) | 5.71 [4.68 to 6.15] | 3.98 [3.48 to 5.69]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.079, Wilcoxon (Mann-Whitney)

44. Secondary Outcome: Osteoid Thickness (OTh.) in the Endocortical Compartment of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: Osteoid thickness (OTh.) in the endocortical compartment is a measure of the average thickness of osteoid seams.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had OTh. analysis of the EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: micrometer (µm)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 29
micrometer (µm)
  6 months (n=23, 29) | 4.94 [4.41 to 5.87] | 3.70 [2.99 to 4.82]
  24 months (n=9, 8) | 5.23 [4.22 to 7.24] | 3.53 [3.21 to 5.07]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — P-value is for 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.039, Wilcoxon (Mann-Whitney) — P-value is for 24 months

45. Secondary Outcome: Wall Thickness (WTh.) in the Cancellous Compartment of Iliac Crest Bone Biopsies at 6 Months
Description: Wall thickness (WTh.) in the cancellous compartment is measured as the mean distance from the cement line to the marrow space of completed trabecular bone packets.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
µm | 31.29 (3.25) [28.80 to 33.26] | 28.63 (2.59) [27.16 to 30.43]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.014, Wilcoxon (Mann-Whitney)

46. Secondary Outcome: Wall Thickness (WTh.) in the Cancellous Compartment of Iliac Crest Bone Biopsies at 24 Months
Description: as for outcome 45
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had WTh. analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: micrometer (µm)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 9
micrometer (µm) | 31.37 [28.29 to 32.34] | 29.26 [27.04 to 29.66]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.079, Wilcoxon (Mann-Whitney)

47. Secondary Outcome: Wall Thickness (WTh.) in the Endocortical Compartment of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: Wall thickness (WTh.) in the endocortical compartment is measured as the mean distance from the cement line to the marrow space of completed trabecular bone packets.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had WTh. analysis of the EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: micrometer (µm)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 29
micrometer (µm)
  6 months (n=23, 29) | 36.30 [34.27 to 37.62] | 32.39 [29.45 to 36.20]
  24 months (n=9, 8) | 34.00 [33.59 to 36.92] | 32.45 [31.43 to 36.44]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.027, Wilcoxon (Mann-Whitney) — P-value is for 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.268, Wilcoxon (Mann-Whitney) — P-value is for 24 months

48. Secondary Outcome: Percentage of Eroded Surface/Bone Surface (ES/BS) in the Cancellous Compartment of Iliac Crest Bone Biopsies at 6 Months
Description: Eroded surface/bone surface (ES/BS) in the cancellous compartment is the fraction of the entire trabecular surface occupied by resorption bays, including both those with and without osteoclasts. It is an indicator of bone resorption.
Time Frame: 6 months
Population: All randomized participants who received at least one dose of study drug with an evaluable bone biopsy.
Measure: Median (Inter-Quartile Range); unit: percentage of surface
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 28 | 30
percentage of surface | 4.59 [3.14 to 6.01] | 2.71 [1.73 to 3.21]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

49. Secondary Outcome: Percentage of Eroded Surface/Bone Surface (ES/BS) in the Cancellous Compartment of Iliac Crest Bone Biopsies at 24 Months
Description: as for outcome 48
Time Frame: 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had ES/BS analysis of the CC at 24 months.
Measure: Median (Inter-Quartile Range); unit: percentage of surface
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 10 | 9
percentage of surface | 4.44 [4.02 to 6.16] | 2.39 [1.87 to 3.66]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.025, Wilcoxon (Mann-Whitney)

50. Secondary Outcome: Percentage of Eroded Surface/Bone Surface (ES/BS) in the Endocortical Compartment of Iliac Crest Bone Biopsies at 6 and 24 Months
Description: Eroded surface/bone surface (ES/BS) in the endocortical compartment is the fraction of the entire trabecular surface occupied by resorption bays, including both those with and without osteoclasts. It is an indicator of bone resorption.
Time Frame: 6 and 24 months
Population: All participants who received at least one dose of study drug with an evaluable bone biopsy and had ES/BS analysis of the EC at 6 and 24 months.
Measure: Median (Inter-Quartile Range); unit: percentage of surface
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 23 | 29
percentage of surface
  6 months (n=23, 29) | 4.06 [1.92 to 6.32] | 1.87 [1.54 to 3.33]
  24 months (n=9, 8) | 3.43 [2.10 to 4.72] | 1.88 [1.55 to 2.27]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.012, Wilcoxon (Mann-Whitney) — P-value is for 6 months
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p = 0.092, Wilcoxon (Mann-Whitney) — P-value is for 24 months

51. Secondary Outcome: Change From Baseline in Serum Carboxyterminal Cross-Linking Telopeptide of Type I Collagen (CTX) at Month 1, 3 and 6 Endpoint
Description: CTX is a measure of bone resorption.
Time Frame: Baseline, 1, 3, 6 months
Population: All randomized participants who received at least one dose of study drug with available biochemical marker of bone turnover data.
Measure: Median (Inter-Quartile Range); unit: nanogram/milliliter (ng/mL)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 34 | 35
nanogram/milliliter (ng/mL)
  Change at 1 month (n= 32, 31) | 0.06 (0.20) [-0.04 to 0.15] | -0.37 (0.20) [-0.46 to -0.29]
  Change at 3 months (n= 32, 29) | 0.26 (0.35) [0.06 to 0.51] | -0.35 (0.19) [-0.42 to -0.29]
  Change at 6 months (n= 25, 28) | 0.31 (0.48) [0.19 to 0.75] | -0.32 (0.19) [-0.42 to -0.23]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value is for change from baseline at 1 month
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value is for change from baseline at 3 months
Statistical Analysis 3: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value is for change from baseline at 6 months

52. Secondary Outcome: Change From Baseline in Serum Carboxyterminal Cross-Linking Telopeptide of Type I Collagen (CTX) at Month 12 Endpoint
Description: CTX is a measure of bone resorption.
Time Frame: Baseline, 12 months
Population: All participants who received at least one dose of study drug, had baseline and 12 months CTX measurement.
Measure: Median (Inter-Quartile Range); unit: nanogram/milliliter (ng/mL)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 26 | 28
nanogram/milliliter (ng/mL) | 0.42 [0.22 to 0.66] | -0.23 [-0.35 to -0.18]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

53. Secondary Outcome: Change From Baseline in Serum Procollagen Type I N-Terminal Propeptide (PINP) at Month 1, 3 and 6 Endpoint
Description: PINP is a measure of bone formation.
Time Frame: Baseline, 1, 3, 6 months
Population: as for outcome 51
Measure: Median (Inter-Quartile Range); unit: microgram/Liter (µg/L)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 34 | 35
microgram/Liter (µg/L)
  Change at 1 month (n= 32, 31) | 65.50 (32.03) [35.50 to 82.00] | -15.00 (9.27) [-21.00 to -11.00]
  Change at 3 months (n= 32, 29) | 66.00 (68.65) [33.50 to 107.50] | -39.00 (14.58) [-47.00 to -28.00]
  Change at 6 months (n= 25, 28) | 84.00 (135.90) [63.00 to 155.00] | -37.50 (16.44) [-48.50 to -26.50]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value is for change from baseline at 1 month
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value is for change from baseline at 3 months
Statistical Analysis 3: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value is for change from baseline at 6 months

54. Secondary Outcome: Change From Baseline in Serum Procollagen Type I N-Terminal Propeptide (PINP) at Month 12 Endpoint
Description: PINP is a measure of bone formation.
Time Frame: Baseline, 12 months
Population: All participants who received at least one dose of study drug, had baseline and 12 months PINP measurement.
Measure: Median (Inter-Quartile Range); unit: microgram/liter (µg/L)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 26 | 28
microgram/liter (µg/L) | 93.50 [49.00 to 155.00] | -33.00 [-38.00 to -21.50]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

55. Secondary Outcome: Change From Baseline in Serum Osteocalcin (OC) at Month 1, 3, and 6 Endpoint
Description: OC is a measure of osteoblast function.
Time Frame: Baseline, 1, 3, 6 months
Population: as for outcome 51
Measure: Median (Inter-Quartile Range); unit: µg/L
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 34 | 35
µg/L
  Change at 1 month (n= 32, 32) | 22.35 (11.58) [17.89 to 29.01] | -3.39 (2.82) [-4.64 to -1.28]
  Change at 3 months (n=32, 30) | 29.93 (19.02) [20.03 to 40.67] | -12.30 (5.01) [-13.39 to -8.08]
  Change at 6 months (n= 25, 29) | 30.85 (33.21) [22.78 to 56.22] | -14.06 (7.15) [-15.97 to -11.08]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value is for change from baseline at 1 month
Statistical Analysis 2: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value is for change from baseline at 3 months
Statistical Analysis 3: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — P-value is for change from baseline at 6 months

56. Secondary Outcome: Change From Baseline in Serum Osteocalcin (OC) at Month 12 Endpoint
Description: OC is a measure of osteoblast function.
Time Frame: Baseline, 12 months
Population: All participants who received at least one dose of study drug, had baseline and 12 months OC measurements.
Measure: Median (Inter-Quartile Range); unit: microgram/liter (µg/L)
Arm/Group | Teriparatide | Zoledronic Acid
Number analyzed (Participants) | 26 | 30
microgram/liter (µg/L) | 32.98 [15.14 to 45.56] | -12.32 [-15.42 to -8.22]
Statistical Analysis 1: Comparison: Teriparatide vs Zoledronic Acid; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events were updated to add the adverse events that occurred during the 12 month extension period to the adverse events that were previously reported from the initial 12 month period.
Arm/Group | Teriparatide | Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 2/34 | 3/35
Other Adverse Events (participants affected / at risk) | 31/34 | 31/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=34) | Zoledronic Acid (N=35)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=34) | Zoledronic Acid (N=35)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 4 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Chills (General disorders) | 1 (1) | 3 (3)
Cyst (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 2 (3)
Pain (General disorders) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6) | 4 (5)
Sinusitis (Infections and infestations) | 2 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 4 (5)
Procedural pain (Injury, poisoning and procedural complications) | 8 (9) | 9 (10)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 8 (9)
Migraine (Nervous system disorders) | 2 (2) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 4 (4) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days